CLINICAL TRIAL: NCT05914766
Title: PATHWAYS: An Informational and Supportive Care Intervention for Patients With Locally Advanced Rectal Cancer
Brief Title: An Informational and Supportive Care Intervention for Patients With Locally Advanced Rectal Cancer
Acronym: PATHWAYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kelsey S. Lau-Min, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-115
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer; Self Efficacy
Keywords: total neoadjuvant therapy; locally advanced rectal cancer; self efficacy; psychoeducational; multimodality treatment
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention or enhanced usual care. Randomization will be stratified by treatment sequence (e.g., chemotherapy first vs. concurrent chemoradiation first).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study Phase I: PATHWAYS Intervention (Experimental): Participants assigned to the PATHWAYS Intervention will receive: 1) four coaching sessions, 2) a comprehensive patient education guidebook, and 3) a coaching session workbook.
  Interventions: Behavioral: PATHWAYS
- Study Phase I: Enhanced Usual Care (Active Comparator): Participants assigned to the enhanced usual care will receive: 1) an information resource guide for navigating information online.
  Interventions: Other: Enhanced usual care
- Study Phase II: PATHWAYS Intervention (Experimental): Participants assigned to the PATHWAYS Intervention will receive: 1) four coaching sessions and 2) a comprehensive patient education guidebook. The intervention has been modified and refined based on feedback from Study Phase I.
  Interventions: Behavioral: PATHWAYS
- Study Phase II: Enhanced Usual Care (Active Comparator): Participants assigned to the enhanced usual care will receive: 1) an information resource guide for navigating information online.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: PATHWAYS — The PATHWAYS intervention is a psychoeducational intervention comprised of four behavioral coaching sessions and a patient education guidebook.
  Arms: Study Phase I: PATHWAYS Intervention; Study Phase II: PATHWAYS Intervention
Other: Enhanced usual care — The enhanced usual care condition consists of an information resource guide.
  Arms: Study Phase I: Enhanced Usual Care; Study Phase II: Enhanced Usual Care

SUMMARY:
The aim of this study is to evaluate the feasibility and acceptability of conducting a randomized trial of a brief psychoeducational intervention versus enhanced usual care for patients with locally advanced rectal cancer who are initiating neoadjuvant multimodality treatment.

DETAILED DESCRIPTION:
This is a randomized controlled trial that is split into two phases. Study Phase I tested the feasibility and acceptability of a study evaluating a psychoeducational intervention relative to a control condition for improving self-efficacy in patients with locally advanced rectal cancer initiating multimodality treatment. This phase enrolled 20 participants.

Study Part 2 was initially planned as an adequately powered RCT to evaluate intervention efficacy for enhancing patient self-efficacy for managing treatment-related challenges and maintaining quality of life. Due to the substantial refinements that were made to the PATHWAYS intervention and study procedures after Study Part 1, we have elected to change Study Part 2 to a second pilot randomized controlled trial to evaluate the feasibility and acceptability of the refined PATHWAYS study among a larger group of patients (n=60).

Participants in the intervention arm will be invited to receive the PATHWAYS intervention, including 4 coaching sessions with a study clinician focused on information and support related to multimodality treatment for LARC. Participants in the control arm will receive an information resource guide that is tailored for patients with LARC.

It is expected that about 80 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Within 8 weeks after documented decision to pursue multi-modality therapy for newly diagnosed LARC (i.e., stage II or III disease)
3. Able to complete study procedures English or with the assistance of an interpreter

Exclusion Criteria:

1. Comorbid health condition that would interfere with study participation, as identified by cancer care team
2. Has undergone treatment for a prior colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2028-05-21 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants retained in the intervention (feasibility) | 4 weeks
  The primary outcome will be feasibility, defined as ≥60% retention of participants over the four-week intervention.

SECONDARY OUTCOMES:
Proportion of patients enrolled on the study (feasibility) | 12 weeks
  A secondary feasibility outcome will be defined as ≥60% enrollment among all eligible patients
Proportion of participants reporting acceptability of the intervention (acceptability) | 12 weeks
  A secondary outcome of acceptability will be defined as ≥80% of participants in the intervention arm reporting Client Satisfaction Questionnaire (CSQ-8) scores of ≥20 (scale from 8-32, higher scores indicate higher satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Lau-Min, MD, MSCE, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at link below